CLINICAL TRIAL: NCT01615679
Title: Integrated Diagnosis and Treatment of Adults With Attention-deficit/Hyperactivity Disorder (ADHD)
Brief Title: Integrated Diagnosis and Treatment of Adults With Attention-deficit/Hyperactivity Disorder
Acronym: IDEA
Status: Completed | Type: Observational
Sponsor: Medice Arzneimittel Pütter GmbH & Co KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 6520-0660-02
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Adult Attention-deficit/Hyperactivity Disorder
Keywords: Non-interventional study; Attention Deficit/Hyperactivity Disorder; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-interventional study to gain further information about the therapy progression in routine treatment of adults with attention-deficit/hyperactivity disorder (ADHD). Main focus will be on the improvement of the clinical global impression (CGI) in comparison to the outcome of randomized, controlled studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with newly diagnosed ADHD

Exclusion Criteria:

* Known sensitivity to methylphenidate or any of the excipients
* Glaucoma
* Phaeochromocytoma
* During treatment with non-selective, irreversible monoamine oxidase (MAO) inhibitors, or within a minimum of 14 days of discontinuing those drugs, due to risk of hypertensive crisis
* Hyperthyroidism or Thyrotoxicosis
* Diagnosis or history of severe depression, anorexia nervosa/anorexic disorders, suicidal tendencies, psychotic symptoms, severe mood disorders, mania, schizophrenia, psychopathic/borderline personality disorder.
* Diagnosis or history of severe and episodic (Type I) Bipolar (affective) Disorder (that is not well-controlled)
* pre-existing cardiovascular disorders including severe hypertension, heart failure, arterial occlusive disease, angina, haemodynamically significant congenital heart disease, cardiomyopathies, myocardial infarction, potentially life-threatening arrhythmias and channelopathies (disorders caused by the dysfunction of ion channels)
* pre-existing cerebrovascular disorders cerebral aneurysm, vascular abnormalities including vasculitis or stroke
* a history of pronounced anacidity of the stomach with a pH value above 5.5, in therapy with H2-receptor blockers or in antacid therapy,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with newly diagnosed ADHD who shall be treated with Medikinet(R) adult.
Sampling Method: Non-Probability Sample
Enrollment: 468 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression (CGI) | 12-14 weeks

SECONDARY OUTCOMES:
Wender-Reimherr adult attention deficit disorder scale (WRAADDS) - self-report | 12-14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roland Fischer, Dr., Study Chair — Medice Arzneimittel Pütter GmbH & Co KG; Michael Rösler, Prof. Dr., Study Director — Universität des Saarlandes, Institut für Gerichtliche Psychologie und Psychiatrie
Locations (1):
- Universität des Saarlandes, Gerichtliche Psychologie und Psychiatrie, Homburg, Germany